CLINICAL TRIAL: NCT03468855
Title: An Open-Label Pilot Study of the Safety, Tolerability and Efficacy of ATI-50002 Topical Solution Administered Twice-Daily in Adult Subjects With Non-Segmental Facial Vitiligo
Brief Title: A Study of ATI-50002 Topical Solution for the Treatment of Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI-50002-VITI-201
Record Dates: First submitted 2018-02-12; First posted 2018-03-19 (Actual); Results first posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATI-50002 Topical Solution (Experimental): ATI-50002 topical solution, high dose active, twice-daily, 24 weeks
  Interventions: Drug: ATI-50002 topical solution

INTERVENTIONS:
Drug: ATI-50002 topical solution — Topical Solution administered twice daily

SUMMARY:
The main objective of this study is to assess the safety, tolerability and efficacy of ATI-50002 Topical Solution, 0.46% in subjects with non-segmental facial vitiligo.

DETAILED DESCRIPTION:
This is a multicenter, open-label study designed to evaluate the safety, tolerability and efficacy of ATI-50002 Topical Solution 0.46% in subjects with non-segmental facial vitiligo. Subjects will be required to have a clinical diagnosis of non-segmental facial vitiligo effecting at least 0.25% of total body surface area (TBSA) (excluding upper and lower eyelids, mucosal lip areas, and forehead and chin areas covered by the stereotactic positioning device for photography) with at least one area of the face with normal pigmentation. Twenty-four eligible subjects will receive ATI-50002 Topical Solution, 0.46%, BID for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a clinical diagnosis of new onset or actively progressing non-segmental facial vitiligo or worsening of existing facial lesions within the past 6 months.
2. Subject has non-segmental facial vitiligo effecting at least 0.25% total body surface area (TBSA) (excluding the upper and lower eyelids, mucosal lip areas and forehead and chin areas covered by the stereotactic positioning device for photography) with at least one area of the face with normal pigmentation.
3. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at the baseline visit and must agree to use an approved method of highly effective birth control for the duration of the study and for 30 days after last study medication application.
4. Subject is in good general health and free of any known disease state or physical condition which, in the opinion of the investigator, would interfere with the study assessments or put the subject at undue risk by study participation.
5. Subject agrees to refrain from any other treatments for vitiligo from the screening visit through the final follow-up visit. Over the counter (OTC) preparations deemed acceptable by the investigator and camouflage makeups are permitted.

Exclusion Criteria:

1. Subject with evidence of poliosis (white hairs) in > 50% of their facial vitiligo lesions.
2. Subject with total facial depigmentation.
3. Subject with spontaneous ongoing repigmentation (documented based on the subject's reporting in the last 3 months).
4. Subject who has segmental vitiligo.
5. Subject who has failed phototherapy. Failed phototherapy is defined as failure to achieve satisfactory repigmentation following adequately delivered phototherapy as determined by the investigator.
6. Subject currently has, or has a history of, skin disease (e.g., psoriasis, seborrheic dermatitis, etc.) that, in the opinion of the investigator, would interfere with the study medication application or study assessments.
7. Subject has, or has a history of, severe, progressive or uncontrolled autoimmune, metabolic, renal, hepatic, gastrointestinal, pulmonary, cardiovascular, genitourinary (i.e.,renal disease), hematological disease, neurologic or cerebral disorders, infectious disease or coagulation disorders that, in the opinion of the investigator, would interfere with the study assessments or put the subject at undue risk by study participation.
8. Subject currently has a history of, current, or suspected systemic or cutaneous malignancy and/or lymphoproliferative disease, other than a history of adequately treated, well healed and completely cleared non-melanoma skin cancers (e.g., basal or squamous cell carcinoma) treated successfully at least 1 year prior to study entry with no evidence of disease.
9. Subject currently has evidence of active or latent bacterial (including tuberculosis) or viral infections at the time of enrollment, or a history of incompletely treated or untreated tuberculosis. Subjects who have initiated therapy for latent tuberculosis for at least 2 weeks and agree to continue their therapy through completion may participate.
10. Subject has a history of serious local infection (e.g., cellulitis, abscess) or systemic infection, or history of treated infection (e.g., pneumonia, septicemia) within 3 months prior to the baseline visit. Subjects on an antibiotic for a nonserious, acute local infection must complete the course prior to enrollment into the study.
11. Subject has herpes zoster or cytomegalovirus (CMV) that resolved within 8 weeks prior to Visit 1.
12. Subject has a history of frequent outbreaks of oral Herpes Simplex Virus defined as more than 4 episodes per year.
13. Subjects previously treated with depigmenting agents.
14. Clinically significant laboratory abnormalities at screening that in the opinion of the investigator, would make the subject a poor candidate for the study.
15. Subject who has an absolute neutrophil count <1,000/mm3, or platelet count < 50,000/mL.
16. Subject unable to comply with the required washout periods
17. Subject who has participated in any investigational drug or device trial, regardless of indication in which administration of an investigational drug or device occurred within 30 days or 5 half-lives (whichever is longer) of screening (Visit 1). Note that investigational treatment for vitiligo (in any body area) requires a longer washout
18. Subjects with a clinically significant abnormal thyroid-stimulating hormone or free T4 at screening. Subjects under treatment with stable thyroid replacement who have a free T4 and TSH within the normal range may participate.
19. Subject has history of sensitivity to any of the ingredients in the study medication.
20. Subject has a history of, or current alcohol or drug abuse within 2 years of study enrollment.
21. Screening ECG findings of:

    1. QTcF >450msec for males or >470msec for females (use of the ECG algorithm is acceptable for this purpose)
    2. Heart rate ≤ 45 or ≥ 100 beats/minutes
    3. Rhythm disturbance other than sinus arrhythmia or ectopic supraventricular rhythm (ectopic atrial rhythm)
    4. Conduction disturbance including PR >240msec, pre-excitation (delta wave and PR <120msec), second degree or higher AV block
    5. Acute or chronic signs of ischemia.
    6. Left Bundle Branch Block
    7. Prior myocardial infarction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Aclaris Investigator Site, Encinitas, California
  - Aclaris Investigator Site, Los Angeles, California
  - Aclaris Investigator Site, Worcester, Massachusetts
  - Aclaris Investigator Site, Dallas, Texas
  - Aclaris Investigator Site, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ATI-50002 0.46% Topical Solution: ATI-50002 0.46% topical solution, high dose active, twice-daily, 24 weeks
  ATI-50002 0.46% topical solution: Topical Solution administered twice daily
Period: Overall Study
Arm/Group | ATI-50002 0.46% Topical Solution
Started | 34
Completed | 23
Not Completed | 11
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 3
Not completed — Inclusion/Exclusion Enrollment Violator | 1

BASELINE CHARACTERISTICS:
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 27
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 34
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I - Always Burns | 0
  II - Burns Easily | 5
  III - Burns Moderately | 16
  IV - Burns Minimally | 9
  V - Rarely Burns | 3
  VI - Never Burns | 1
Duration of Vitiligo Disease (years) (n) [Mean (Standard Deviation); unit: years] | 13.6 (10.47)
Duration of Current Episode (years) (n) [Mean (Standard Deviation); unit: years] | 3.9 (7.24)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Facial Depigmentation in the AOI (Area of Interest) Based on Canfield 2-D Photographic Analysis From Baseline to Week 24
Description: Mean change from baseline in facial depigmentation in quantified Area of Interest (AOI) using Canfield-2-D photographic image analysis from baseline (Visit 2) compared to Week 24. Facial depigmentation is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 24 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
score on a scale | 2.0 (8.41)

2. Secondary Outcome: Mean Change From Baseline in Facial Depigmentation in the AOI (Area of Interest) Based on Canfield 2-D Photographic Analysis From Baseline Compared to Week 48
Description: Mean change from baseline in facial depigmentation in quantified Area of Interest (AOI) using Canfield-2-D photographic image analysis from baseline (Visit 2) compared to Week 48. Facial depigmentation is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 48 Weeks
Population: Subjects completing 24 weeks of treatment have the option to extend treatment for an additional 24 weeks. Subjects not wishing to continue treatment can withdraw consent.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 16
score on a scale | -1.4 (15.11)

3. Secondary Outcome: Mean Change From Baseline in Facial Depigmentation in the AOI (Area of Interest) Based on Canfield 2-D Photographic Analysis From Baseline Compared to Week 4
Description: Mean change from baseline in facial depigmentation in quantified Area of Interest (AOI) using Canfield-2-D photographic image analysis from baseline (Visit 2) compared to Week 4. Facial depigmentation is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 4 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
score on a scale | 0.2 (4.47)

4. Secondary Outcome: Mean Change From Baseline in Facial Depigmentation in the AOI (Area of Interest) Based on Canfield 2-D Photographic Analysis From Baseline Compared to Week 8
Description: Mean change from baseline in facial depigmentation in quantified Area of Interest (AOI) using Canfield-2-D photographic image analysis from baseline (Visit 2) compared to Week 8. Facial depigmentation is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
score on a scale | 0.5 (4.82)

5. Secondary Outcome: Mean Change From Baseline in Facial Depigmentation in the AOI (Area of Interest) Based on Canfield 2-D Photographic Analysis From Baseline Compared to Week 12
Description: Mean change from baseline in facial depigmentation in quantified Area of Interest (AOI) using Canfield-2-D photographic image analysis from baseline (Visit 2) compared to Week 12. Facial depigmentation is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 12 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
score on a scale | 0.3 (9.04)

6. Secondary Outcome: Mean Change From Baseline in Facial Depigmentation in the AOI (Area of Interest) Based on Canfield 2-D Photographic Analysis From Baseline Compared to Week 16
Description: as for outcome 3
Time Frame: Baseline to 16 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
score on a scale | -0.8 (8.20)

7. Secondary Outcome: Mean Change From Baseline in Facial Depigmentation in the AOI (Area of Interest) Based on Canfield 2-D Photographic Analysis From Visit 2 Compared to Week 20
Description: Mean change from baseline in facial depigmentation in quantified Area of Interest (AOI) using Canfield-2-D photographic image analysis from baseline (Visit 2) compared to Week 20. Facial depigmentation is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 20 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
score on a scale | 1.3 (9.22)

8. Secondary Outcome: Mean Change From Baseline in Facial Depigmentation in the AOI (Area of Interest) Based on Canfield 2-D Photographic Analysis From Baseline Compared to Week 32
Description: as for outcome 3
Time Frame: Baseline to 32 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 16
score on a scale | 4.2 (9.09)

9. Secondary Outcome: Mean Change From Baseline in Facial Depigmentation in the AOI (Area of Interest) Based on Canfield 2-D Photographic Analysis From Baseline Compared to Week 40
Description: Mean change from baseline in facial depigmentation in quantified Area of Interest (AOI) using Canfield-2-D photographic image analysis from baseline (Visit 2) compared to Week 40. Facial depigmentation is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 40 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 16
score on a scale | 1.9 (12.14)

10. Secondary Outcome: Mean Change From Baseline in Facial Depigmentation in the AOI (Area of Interest) Based on Canfield 2-D Photographic Analysis From Baseline Compared to Post-treatment Week 52
Description: Mean change from baseline in facial depigmentation in quantified Area of Interest (AOI) using Canfield-2-D photographic image analysis from baseline (Visit 2) compared to Week 52. Facial depigmentation is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 16
score on a scale | -1.4 (13.29)

11. Secondary Outcome: Mean Change From Baseline in the Facial Assessment of the Vitiligo Area Scoring Index (F-VASI) Compared to Week 4
Description: The Facial Vitiligo Area Scoring Index (F-VASI) is an assessment of the subject's facial vitiligo modified from the Vitiligo Area Scoring Index for the face only at week 4. F-VASI is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 4 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
score on a scale | -0.023 (0.0946)

12. Secondary Outcome: Mean Change From Baseline in the Facial Assessment of the Vitiligo Area Scoring Index (F-VASI) Compared to Week 8
Description: The Facial Vitiligo Area Scoring Index (F-VASI) is an assessment of the subject's facial vitiligo modified from the Vitiligo Area Scoring Index for the face only at Week 8. F-VASI is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
score on a scale | -0.043 (0.1454)

13. Secondary Outcome: Mean Change From Baseline in the Facial Assessment of the Vitiligo Area Scoring Index (F-VASI) Compared to Week 12
Description: The Facial Vitiligo Area Scoring Index (F-VASI) is an assessment of the subject's facial vitiligo modified from the Vitiligo Area Scoring Index for the face only at week 12. F-VASI is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 12 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
score on a scale | -0.071 (0.2049)

14. Secondary Outcome: Mean Change From Baseline in the Facial Assessment of the Vitiligo Area Scoring Index (F-VASI) Compared to Week 16
Description: The Facial Vitiligo Area Scoring Index (F-VASI) is an assessment of the subject's facial vitiligo modified from the Vitiligo Area Scoring Index for the face only at week 16. F-VASI is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
score on a scale | -0.065 (0.2116)

15. Secondary Outcome: Mean Change From Baseline in the Facial Assessment of the Vitiligo Area Scoring Index (F-VASI) Compared to Week 20
Description: The Facial Vitiligo Area Scoring Index (F-VASI) is an assessment of the subject's facial vitiligo modified from the Vitiligo Area Scoring Index for the face only at week 20. F-VASI is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 20 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
score on a scale | -0.070 (0.2063)

16. Secondary Outcome: Mean Change From Baseline in the Facial Assessment of the Vitiligo Area Scoring Index (F-VASI) Compared to Week 24
Description: The Facial Vitiligo Area Scoring Index (F-VASI) is an assessment of the subject's facial vitiligo modified from the Vitiligo Area Scoring Index for the face only at week 24. F-VASI is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 24 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
score on a scale | -0.067 (0.2411)

17. Secondary Outcome: Mean Change From Baseline in the Facial Assessment of the Vitiligo Area Scoring Index (F-VASI) Compared to Week 32
Description: The Facial Vitiligo Area Scoring Index (F-VASI) is an assessment of the subject's facial vitiligo modified from the Vitiligo Area Scoring Index for the face only at week 32. F-VASI is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 32 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 16
score on a scale | -0.004 (0.1945)

18. Secondary Outcome: Mean Change From Baseline in the Facial Assessment of the Vitiligo Area Scoring Index (F-VASI) Compared to Week 40
Description: The Facial Vitiligo Area Scoring Index (F-VASI) is an assessment of the subject's facial vitiligo modified from the Vitiligo Area Scoring Index for the face only at week 40. F-VASI is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 40 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 16
score on a scale | -0.076 (0.3567)

19. Secondary Outcome: Mean Change From Baseline in the Facial Assessment of the Vitiligo Area Scoring Index (F-VASI) Compared to Week 48
Description: The Facial Vitiligo Area Scoring Index (F-VASI) is an assessment of the subject's facial vitiligo modified from the Vitiligo Area Scoring Index for the face only at week 48. F-VASI is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 48 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 16
score on a scale | -0.121 (0.4062)

20. Secondary Outcome: Mean Change From Baseline in the Facial Assessment of the Vitiligo Area Scoring Index (F-VASI) Compared to Post-treatment Week 52
Description: The Facial Vitiligo Area Scoring Index (F-VASI) is an assessment of the subject's facial vitiligo modified from the Vitiligo Area Scoring Index for the face only at week 52. F-VASI is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 16
score on a scale | -0.158 (0.4785)

21. Secondary Outcome: Treatment Success Based on the Subject's Assessment of Vitiligo on the Vitiligo Noticeability Scale (VNS) at Week 4
Description: The Vitiligo Noticeability Scale (VNS) represents the subject's assessment of the noticeability of facial vitiligo during the study treatment period by means of answering the question, "Compared to before treatment, how noticeable is the vitiligo now?" Subject response options include, "1: More Noticeable", "2: As Noticeable", "3: Slightly Less Noticeable", "4: A Lot Less Noticeable", and "5: No Longer Noticeable". Treatment success will be defined as follows: VNS score of 1 or 2 = treatment not successful, VNS score of 3 = treatment partially successful, or VNS score of 4 or 5 = treatment successful. Higher scores represent better outcomes.
Time Frame: Baseline to 4 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 29
score on a scale | 2.1 (0.58)

22. Secondary Outcome: Treatment Success Based on the Subject's Assessment of Vitiligo on the Vitiligo Noticeability Scale (VNS) at Week 8
Description: as for outcome 21
Time Frame: Baseline to 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 27
score on a scale | 2.1 (0.58)

23. Secondary Outcome: Treatment Success Based on the Subject's Assessment of Vitiligo on the Vitiligo Noticeability Scale (VNS) at Week 12
Description: as for outcome 21
Time Frame: Baseline to 12 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 27
score on a scale | 2.1 (0.68)

24. Secondary Outcome: Treatment Success Based on the Subject's Assessment of Vitiligo on the Vitiligo Noticeability Scale (VNS) at Week 16
Description: as for outcome 21
Time Frame: Baseline to 16 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 25
score on a scale | 2.1 (0.67)

25. Secondary Outcome: Treatment Success Based on the Subject's Assessment of Vitiligo on the Vitiligo Noticeability Scale (VNS) at Week 20
Description: as for outcome 21
Time Frame: Baseline to 20 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 24
score on a scale | 2.3 (0.53)

26. Secondary Outcome: Treatment Success Based on the Subject's Assessment of Vitiligo on the Vitiligo Noticeability Scale (VNS) at Week 24
Description: as for outcome 21
Time Frame: Baseline to 24 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 24
score on a scale | 2.2 (0.66)

27. Secondary Outcome: Treatment Success Based on the Subject's Assessment of Vitiligo on the Vitiligo Noticeability Scale (VNS) at Week 32
Description: as for outcome 21
Time Frame: Baseline to 32 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 14
score on a scale | 2.1 (0.73)

28. Secondary Outcome: Treatment Success Based on the Subject's Assessment of Vitiligo on the Vitiligo Noticeability Scale (VNS) at Week 40
Description: as for outcome 21
Time Frame: Baseline to 40 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 14
score on a scale | 2.4 (0.74)

29. Secondary Outcome: Treatment Success Based on the Subject's Assessment of Vitiligo on the Vitiligo Noticeability Scale (VNS) at Week 48
Description: as for outcome 21
Time Frame: Baseline to 48 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 14
score on a scale | 2.4 (1.01)

30. Secondary Outcome: Mean Change From Baseline in Total VASI at Week 24
Description: The Vitiligo Area Scoring Index (VASI) is an assessment of the subject's Vitiligo Area Scoring Index. VASI is measured on a scale of 0 to 100, with a score of 0 meaning no depigmentation and a score of 100 meaning total depigmentation. Lower scores represent better outcomes.
Time Frame: Baseline to 24 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
score on a scale | 0.340 (1.4829)

31. Secondary Outcome: Mean Change From Baseline in Total VASI at Week 48
Description: as for outcome 30
Time Frame: Baseline to 48 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 34
score on a scale | 0.008 (1.5341)

ADVERSE EVENTS:
Time Frame: The analysis included all treatment-emergent adverse events (TEAEs), defined as any recorded AE that occurred on or after the initiation of study medication and continue reporting until the end of the subject's last study visit (4-week post-treatment follow up visit).
Arm/Group | ATI-50002 0.46% Topical Solution
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 2/34
Other Adverse Events (participants affected / at risk) | 23/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATI-50002 0.46% Topical Solution (N=34)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATI-50002 0.46% Topical Solution (N=34)
Coronary artery disease (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Application site acne (General disorders) | 2 (3)
Application site discolouration (General disorders) | 1 (1)
Application site dryness (General disorders) | 6 (7)
Application site pain (General disorders) | 1 (1)
Application site rash (General disorders) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (6)
Oral herpes (Infections and infestations) | 1 (2)
Pharyngitis (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood pressure systolic increased (Investigations) | 1 (1)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1)
Blood urine present (Investigations) | 2 (2)
Eosinophil count increased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Low density lipoprotein increased (Investigations) | 2 (4)
Protein urine present (Investigations) | 1 (1)
Red blood cell count increased (Investigations) | 1 (1)
Specific gravity urine decreased (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Excessive exercise (Social circumstances) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT03468855/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT03468855/ICF_002.pdf